CLINICAL TRIAL: NCT00748371
Title: Loss of Effect of Aspirin on Platelet Aggregation During Chronic Administration
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding issue
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Oates, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GM15431-JAO1
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Platelet Aggregation
Keywords: platelet aggregation; granule secretion; thromboxane production; prostacyclin production
MeSH Terms: interventions — Aspirin; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): ASA 40mg daily for 8 weeks followed by 3 weeks of observation
  Interventions: Drug: aspirin
- 2 (Experimental): ASA 1300mg daily for 8 weeks followed by 3 weeks of observation
  Interventions: Drug: aspirin
- 3 (Placebo Comparator): Placebo: one Avicel (cellulose) capsule by mouth twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aspirin — 40mg aspirin: one 40-mg aspirin capsule by mouth each morning + one Avicel capsule by mouth each evening
  Other Names: acetylsalicylic acid; ASA
  Arms: 1
Drug: aspirin — 1300mg aspirin: one 650-mg capsule by mouth twice daily
  Other Names: acetylsalicylic acid; ASA
  Arms: 2
Drug: placebo — Placebo: one Avicel (cellulose) capsule by mouth twice daily
  Other Names: Avicel; cellulose
  Arms: 3

SUMMARY:
Aspirin has shown to be beneficial to some patients with certain diseases such as coronary artery disease or stroke. We are investigating how aspirin works on regulating platelets and thromboxane over time at different doses. We hope to find the best dose of aspirin and/or other medications to help people who are at risk for heart attack or stroke.

DETAILED DESCRIPTION:
he purpose of the study is to better understand the mechanism for failure of daily aspirin administration to prevent cardiovascular events in some at risk individuals. We seek to describe the effect of chronic aspirin administration at varying doses on platelet aggregation. This will help to define mechanisms for aspirin failure and to pursue possible alternative therapies in patients who fail to respond to aspirin therapy.

We hypothesize that (1) inhibition by aspirin (ASA) of ex vivo-induced platelet aggregation varies in a predictable time and dose dependent manner, (2) thromboxane and prostacyclin production is inhibited by ASA in a dose-dependent manner and remains relatively constant over time once maximal inhibition has occurred, and (3) granule secretion by platelets during induced aggregation is inhibited by aspirin acutely but this effect does not persist during chronic administration at high doses.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age 18-40 years
* Non-smokers

Exclusion Criteria:

* ASA/NSAID use previous 14 days.
* Evidence of ASA/NSAID use within previous 14 days at baseline visit based on investigator interpretation of platelet aggregation and platelet secretion studies.
* History of chronic NSAID use.
* Currently taking NSAIDs, corticosteroids, or anticoagulants.
* History of coronary artery disease, myocardial infarction, coronary artery bypass grafting, percutaneous angioplasty, diabetes mellitus or stroke.
* History of gastric,duodenal, or esophageal ulcers or serious gastrointestinal bleed.
* History of frequent headaches, pain syndrome, or other condition requiring frequent use of analgesics.
* History of adverse reaction to ASA.
* Initial platelet count <100K/µl or >500K/µl.
* Initial hematocrit <35% or >50%.
* Weight less than 110 pounds.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Comparison of platelet aggregation, serum thromboxane B2 (TxB2) levels, urinary thromboxane metabolite (Tx-M) levels, and urinary prostacyclin metabolite (PGI-M) levels over time and across dose ranges. | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A Oates, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No